CLINICAL TRIAL: NCT00390936
Title: Phase I Multiple Ascending Dose Study to Determine the Safety, Pharmacokinetics and Pharmacodynamics of BMS-582664 in Japanese Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Study of BMS-582664 in Patients With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA182-012
Record Dates: First submitted 2006-10-20; First posted 2006-10-23 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2010-03

CONDITIONS: Solid Tumors
MeSH Terms: interventions — brivanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (No Intervention): 4 dosages
  Interventions: Drug: Brivanib

INTERVENTIONS:
Drug: Brivanib — Tablet, Oral, Brivanib 300 mg, 600 mg, 800 mg, 1000 mg, once daily (cycle 1: Day 1, Day 8 - 35), more than 5 weeks depending on response/toxicity
  Other Names: BMS-582664

SUMMARY:
The purpose of this study is to assess the dose limiting toxicity (DLT) of BMS-582664 and the maximum tolerated dose(MTD) in subjects with advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have measurable disease
* Documented failure to standard therapies exist, or which are determined to be inappropriate by the investigator
* ECOG PS: 0-1

Exclusion Criteria:

* Subjects with centrally located squamous cell carcinoma of the lung

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | at the end of the first cycle of the study
Maximum Tolerated Dose | at the end of the first cycle of the study

SECONDARY OUTCOMES:
To assess any preliminary evidence of anti-tumor activity observed with BMS-582664 | at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol Myers
Locations (1):
- Local Institution, Sunto-Gun, Shizuoka, Japan

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx